CLINICAL TRIAL: NCT07200843
Title: An Investigation of Heel Rise Test, Postural and Tibial Sway During Single-Leg Stance in Pes Planus
Brief Title: Comparison of Lower Extremity Biomechanics and Postural Stability in Individuals With Pes Planus
Status: Completed | Type: Observational
Sponsor: sevilay seda bas (Other)
Responsible Party: Sponsor-Investigator, sevilay seda bas, Asst. Prof., Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: : 2022-08
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pes Planus Group: Participants aged 18 years and older with a navicular drop test result of at least 10 mm were included. Individuals with chronic diseases, hearing or vision impairments, orthopedic injuries or surgical history, and leg length discrepancy were excluded.
  Interventions: Other: Heel rise test and postural/tibial sway measurement

INTERVENTIONS:
Other: Heel rise test and postural/tibial sway measurement — Participants undergo a heel rise test to assess plantar flexor muscle endurance. Postural and tibial sway are measured during single-leg stance using a wearable sensor under eyes-open and eyes-closed conditions. No therapeutic intervention is applied.

SUMMARY:
The goal of this observational study is to examine the relationship between plantar flexor endurance and postural and tibial sway in adults (≥18 years) with pes planus (flatfoot). The main questions it aims to answer are:

Is there a correlation between plantar flexor endurance, postural sway and tibial sway during single-leg stance?

Participants will:

Perform a heel rise test to assess plantar flexor endurance

Stand on one leg while wearing a motion sensor to measure postural and tibial sway

Complete the tests under both eyes-open and eyes-closed conditions

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older
* A navicular drop test result of at least 10 mm

Exclusion Criteria:

* Individuals with chronic diseases, hearing or vision impairments, orthopedic injuries or surgical history, and leg length discrepancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years and older with a navicular drop test result of at least 10 mm. Participants were recruited through convenience sampling from the university student population. Individuals with chronic diseases, hearing or vision impairments, orthopedic injuries or surgical history, or leg length discrepancy were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Plantar flexor endurance measured by heel rise test | Measured once at baseline during the study visit.
  The number of repetitions participants can perform during the heel rise test, assessing the endurance of the plantar flexor muscles. Participants stood on one leg and raised their heels in time with a metronome set at 40 beats per minute. The test ended when the participant was fatigued or unable to continue, and the number of heel rises completed was recorded. The test was performed on both lower limbs.

SECONDARY OUTCOMES:
Postural sway during single-leg stance | Measured once at baseline during the study visit.
  Postural sway was assessed using the Alda Balance Gear wearable sensor. Sensor was assessed for medio-lateral (ML) and antero-posterior (AP) sway. The sensor was placed at the L3-L5 vertebral level using a belt device. Participants performed a single-leg stance for up to 30 seconds under eyes-open (EO) and eyes-closed (EC) conditions. The test ended if balance was lost and the foot touched the ground. Postural sway was recorded only on the dominant limb.
Tibial sway during single-leg stance | Measured once at baseline during the study visit.
  Tibial sway was assessed using the Alda Balance Gear wearable sensor. Sensor was assessed AP and ML sway. The sensor was placed one-third distal on the lower leg. Participants performed a single-leg stance for up to 30 seconds under eyes-open (EO) and eyes-closed (EC) conditions. The test ended if balance was lost and the foot touched the ground. Tibial sway was measured on both lower limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No